CLINICAL TRIAL: NCT00969176
Title: Single and Multiple Dose Trial to Evaluate Pharmacokinetics, -Dynamics and Safety of iv Paracetamol in Preterm and Term Neonates
Brief Title: Pharmacokinetics, -Dynamics and Safety of Intravenous Paracetamol in Neonates
Acronym: PARANEO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Allegaert Karel, University Hospitals Leuven, Belgium
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S51597; EUdraCT nr 2009-011243-39
Record Dates: First submitted 2009-08-27; First posted 2009-09-01 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-12

CONDITIONS: Pain; Fever
Keywords: pain; fever; neonate; preterm; term; newborn
MeSH Terms: conditions — Pain; Fever; Premature Birth | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- paracetamol (No Intervention): not applicable, since all included cases will receive intravenous paracetamol
  Interventions: Drug: paracetamol

INTERVENTIONS:
Drug: paracetamol — Intravenous paracetamol administration in neonates, loading dose 20 mg/kg, followed by a Gestational age-dependent maintenance dose of 10-20 mg/kg/24 h, divided in 4 doses (each 6h)
  Other Names: perfusalgan, perfalgan, paracetamol sintetica

SUMMARY:
The purpose of this study is triple, i.e. document single dose pharmacokinetics and -dynamics of intravenous paracetamol in preterm and term neonates after a loading dose (20 mg/kg iv bolus paracetamol), document multiple dose pharmacokinetics and -dynamics of intravenous paracetamol in preterm and term neonates, based on the daily doses routinely used within the neonatal intensive care unit and as reported in literature. Finally, document safety of single and repeated dose of intravenous paracetamol in preterm and term neonates.

DETAILED DESCRIPTION:
Prospective, single center, open label study on the pharmacokinetics, -dynamics and safety of intravenous paracetamol in preterm and term neonates admitted in the neonatal intensive care unit, University Hospitals Leuven, Belgium. Patients will be included in this study after formal written informed consent of the parent(s). If a painful procedure is anticipated (e.g. surgery), parents should be informed preferably at least 24 h before the clinical indication will appear. Sixty neonates (i.e. < 29 days of postnatal age), either preterm (< 37 weeks gestational age) or term neonates will be included. At least 24 will be preterm neonates in order to ensure that the evaluated population reflects the typical population taken care for at the unit and in order to comply with the suggestions of EMEA (EMEA/CHMP/18922/05). The decision to prescribe paracetamol will be made by the attending neonatologist and in line with the current standing orders in the unit, i.e. either as a monotherapy for mild to moderate pain, independent of the cause (either postoperative, traumatic or medical) of pain or as part of multimodal analgesia for severe pain.

Before initiation of treatment and during any analgesic treatment, prospective evaluation of pain based on a validated and implemented pain scale (Leuven Neonatal Pain Scale, LNPS, Eur J Clin Pharmacol, 2003) is performed to further titrate treatment as needed. Additional administration or adaptation of any other analgesics as well as other concomitant medications will be recorded.

Paracetamol will be administered by either peripheral venous access or by deep venous catheter, ensuring that the study drug will always be administered alone and will be followed by an appropriate flush of normal saline, in line with the current guidelines at the unit. As soon as clinically feasible, the route of administration will be changed from intravenous to either oral (preferred) or rectal administration in line with the guidelines in the unit Plasma samples will be collected through an arterial line if present for clinical needs. In neonates without arterial access, plasma samples will only be collected when venipuncture is performed for clinical indications. The assessment of plasma pharmacokinetics will be based on a population pharmacokinetic approach in line with the EMEA guidelines on pharmacokinetic study in preterm and term neonates. The Leuven unit has published experience with such an approach (Eur J Clin Pharmacol, 2004) in the assessment of propacetamol pharmacokinetics.

Based on this population PK approach, we will focus on both early sampling (distribution volume, loading dose) and late sampling (clearance) while the total blood volume collected will not exceed 1.8 mL/kg for the complete study in line with the guidelines of EMEA on clinical research in children (EMEA website). It is a standing order at the unit that the procedural pain related to venous puncture is routinely treated with oral glucose (30 %).

When feasible, urine collections will be simultaneously performed (urinary bladder catheter in place for clinical indications, or by Uricol collection bag) in order to document aspects of paracetamol metabolism in neonates based on renal clearance in line with earlier studies reported on the assessment of paracetamol metabolism in early life (Acta Pediatric 2005). We anticipate urine collection in at least 20 neonates, of whom at least 8 preterm neonates.

We hereby have the intention to collect data on both pharmacokinetics, metabolism and pharmacodynamics of this drug in neonates.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication of IV administration of paracetamol in neonates, as evaluated by the attending neonatologist

Exclusion Criteria:

* Recent administration of paracetamol (< 48 h) or clinical contra-indication for administration of paracetamol (hepatic failure).

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of intravenous paracetamol in neonates | during administration of iv paracetamol and up to 24 hours after last administration

SECONDARY OUTCOMES:
Pharmacodynamics of intravenous paracetamol in neonates | during administration of iv paracetamol and up to 6 hours after the last administration
Safety of intravenous paracetamol in neonates | during and up to 48 h after last intravenous administration

CONTACTS AND LOCATIONS:
Overall Officials: karel allegaert, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Allegaert K, Naulaers G, Vanhaesebrouck S, Anderson BJ. The paracetamol concentration-effect relation in neonates. Paediatr Anaesth. 2013 Jan;23(1):45-50. doi: 10.1111/pan.12076. Epub 2012 Nov 21. PMID 23170854